CLINICAL TRIAL: NCT06541418
Title: The Effect of Transtheoretical Model Based Behavior Exchange Program on Risky Behaviors of University Students Receiving Health Education
Brief Title: The Effect of Behavior Exchange Program on Risky Behaviors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Collaborators: Medipol University (Other)
Responsible Party: Principal Investigator, Gülşah KÖRPE, Principal Investigator, Istanbul Medipol University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: GUL121312
Record Dates: First submitted 2022-02-22; First posted 2024-08-07 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Risk Behavior
Keywords: risky behavior; transtheoretical model; behavior change
MeSH Terms: conditions — Risk-Taking

STUDY DESIGN:
Intervention Model Description: randomized controlled trial
Who Masked: Participant
Masking Description: Experimental and control groups were masked in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): As a pre-test, 40 students, who were determined in accordance with the research criteria and assigned to the experimental group, were asked to fill in the Sociodemographic data collection form and SCEÖ.
  Before the planned program, students were sent an e-mail and the program days and times were specified. 4 groups of 10 people were formed. Transtheoretic Model Based Behavior Change Program consisting of 7 sessions was given. At the end of the program, the Risky Behavior Evaluation Scale, which was included in the RSS-ÜF, Behavior Change Stages Short Questionnaire, SEYÖ and Soyodemographic data collection form, was applied again. Follow-up was done with the same measurement tools 3 months after the end of the program.
  Interventions: Behavioral: Transtheoretic Model Based Behavior Change Program
- Control Group (No Intervention): As a pre-test, 40 students who were determined in accordance with the research criteria and assigned to the control group were asked to fill in the Sociodemographic data collection form and SCEÖ. For the posttest and 3-month follow-up, the Risky Behavior Evaluation Scale, which was included in the RSS-ÜF, Behavior Change Stages Short Question Form, SEEÖ and Soyodemographic data collection form, was applied again.
  After the Transtheoretical Model-Based Behavior Change Program given to the experimental group ended, a 1-day training program on changing risky behaviors was applied to the control group in September 2021. All students in the experimental group participated in the program.

INTERVENTIONS:
Behavioral: Transtheoretic Model Based Behavior Change Program — The Behavior Change Program was implemented in 7 sessions of 50 minutes, once a week. Each session in the Behavior Change Program; The warm-up exercise consisted of giving general information about the purpose and the main theme of the session, discussion and feedback on the subject, and the planning of the next week, and a closing process. The Transtheoretic Model Based Behavior Change Program was prepared by the researcher with reference to the behavior change programs in the literature and the elements of the Transtheoretic model.
  Arms: Experimental Group

SUMMARY:
Risky behaviors, which derive their source from features specific to adolescence, may also pose problems in other periods of a person's life and have features that prevent them from becoming responsible adults. These behaviors are defined by Jessor as behaviors that cause personal, social or developmental undesirable consequences and are life-threatening or harmful to health and even actions that can lead to death. Risky behaviors in young people are frequently listed as smoking, alcohol/substance use, nutrition, suicide, school dropout, and destructive behaviors (violence against self/others, etc.). It has been conducted with studies that generally do not take into account the stage of change or accept that all individuals' readiness for behavior change is the same. However, the Transtheoretic Model states that the most appropriate initiatives should be used to facilitate the change in which the individual is at the stage of change. He also states that the initiatives applied without considering the individual's readiness for behavior change develop resistance against behavior change. In this study, it was aimed to determine the effect of the behavior change program prepared based on the transtheoretic model on the risky behaviors of university students receiving health education.

DETAILED DESCRIPTION:
Type of Research This study was planned as a randomized controlled experimental study to determine the effect of the Transtheoretical Model-Based Behavior Change Program applied to university students on the tendency to show risky behavior.

The Universe and Place of the Research The general population of the research will consist of students enrolled in the formal education program at Istanbul Medipol University Faculty of Health Sciences between September 2020 and February 2021. Volunteer students who have Turkish literacy skills, are over 18 years old, do not have major-active psychiatric disease, have a high Risk Behavior Scale-University Form score, and are in the Thinking and Preparation phase of change.

2.3. Sample of the Research Sample size was calculated by power analysis. In the calculation made; Predicting a power value of 0.80 and a level of error of 0.05, it was found that the Risk Behaviors Scale-University Form should be administered to at least 348 people from the general population in order to reach the study population. In the calculation made, it was found appropriate to include 40 students in the experimental group and 40 students in the control group. Assignment will be made to the experimental and control groups by making a probabilistic selection from the study universe. One of participants in the experimental group left the study. The study was completed with 79 participants in total.

Variables of the Study

Independent variables

* Transtheoretic model-based behavior change program
* Group consultancy
* Motivational interview

Dependent Variables

* Risky Behaviors Scale-University Form score average
* Behavior Change Stages Short Questionnaire result
* Self-Efficacy-Efficacy Scale mean score

Research Steps

1. In order to identify the risky students in the study population, the University Form of the Risk Behaviors Scale will be applied to the students of the Faculty of Health Sciences.
2. Students with a high score as a result of the Risk Behaviors Scale-University Form will be determined.
3. The Behavior Change Stages Short Questionnaire will be applied to students with a high risky behavior tendency.
4. Students whose behavior change stages are determined as 'Thinking' and 'Preparation' will be included in the study universe.
5. Assignment will be made to the experimental and control groups by making a random selection from the study universe.
6. The Self-Efficacy-Efficacy Scale will be applied to the experimental and control groups.
7. Transtheoretic Model Based Behavior Change Program (Annex-1) will be applied to the experimental group. The behavior change program includes group counseling and motivational interviews. Short training will be given to the control group to reduce risky behaviors after the study.
8. All measurements of the experimental and control groups will be repeated after the program and 3 months after the end of the program.
9. The data will be statistically analyzed and evaluated.
10. The report will be written.

ELIGIBILITY:
Inclusion Criteria:

* Getting a high score on the Risk Behavior Modification-University Form scale
* Stages of change being Thinking or Preparation,
* Being over the age of 18,
* Not having major-active psychiatric disease,
* Having Turkish literacy skills

Exclusion Criteria:

* students who do not meet the inclusion criteria
* who refused to participate in the study

Ages: 18 Years to 33 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 79 (Actual)
Dates: Start 2020-10-15 (Actual); Primary Completion 2021-04-15 (Actual); Study Completion 2021-07-15 (Actual)

PRIMARY OUTCOMES:
Risky behaviors scale-university form | 1 year
  The scale consists of 60 items and sevendimensions such as; antisocial behaviors, smoking, alcohol use, substance use, suicide tendency, eating habitsand school dropout.
  RDÖUF (RBS-UF) is a Likert-type scale consisting of 60 items and seven dimensions. The five-point scale is answered as "always= 5", "usually= 4", "sometimes= 3", "rarely=2" and "never=1". There is no reverse scored item in the scale. Getting a high score on each dimension indicates a higher level of risk in that dimension.
self-efficacy scale | 1 year
  For each item on the 23-item scale; 1-" drink what I don't know", 2-"describes me a little", 3-"I'm undecided", 4-" me best defines me", S-"describes me very well" is requested. The score given for each item is taken as a basis. But 2,4,5,6,7, 10, 11, 12,14,16,17,18,20,22. items are scored in the opposite direction. So from the scale a minimum of 23 and a maximum of 115 points can be obtained.The increase in the total score obtained from the scale, the individual's self-efficacy-efficacy It means that the perception is at a good level.

CONTACTS AND LOCATIONS:
Overall Officials: Leyla KÜÇÜK, 2, Study Chair — Istanbul Cerrahpaşa University
Locations (1):
- Istanbul Medipol University, Istanbul, Beykoz, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
I can share privately if desired.